CLINICAL TRIAL: NCT05345561
Title: A Prospective, Natural History Study to Assess the Occurrence of HPA-1a Alloimmunization in Women Identified at Higher Risk for Fetal and Neonatal Alloimmune Thrombocytopenia (FNAIT)
Brief Title: Study to Assess the Occurrence of HPA-1a Alloimmunization in Women With Higher Risk for Fetal and Neonatal Alloimmune Thrombocytopenia
Status: Completed | Type: Observational
Sponsor: Rallybio (Industry)
Responsible Party: Sponsor
Other Study IDs: IPA2002
Record Dates: First submitted 2022-04-07; First posted 2022-04-26 (Actual); Last update posted 2025-11-06 (Actual); Status verified 2025-11

CONDITIONS: Fetal and Neonatal Alloimmune Thrombocytopenia
Keywords: Alloimmunization; HPA-1a; Fetal and Neonatal Alloimmune Thrombocytopenia; Neonatal thrombocytopenia; Pregnant women
MeSH Terms: conditions — Thrombocytopenia, Neonatal Alloimmune

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Pregnant women: Women with higher risk of FNAIT
  Interventions: Other: Clinical data collection

INTERVENTIONS:
Other: Clinical data collection — Laboratory tests, Vital assessments, Maternal and fetal genotype testing, Antibodies Testing will be performed.

SUMMARY:
A prospective, non-interventional, natural history study to assess the occurrence of higher FNAIT risk across a broad population of different racial and ethnic characteristics and the occurrence of HPA-1a alloimmunization in these women.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant women (≥ 18 years of age) who have provided informed consent for the study.

Exclusion Criteria:

* Participants with prior history of FNAIT

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes
Study Population: Pregnant women presenting at a Gestation Week 10 to 14 pre-natal visit
Sampling Method: Non-Probability Sample
Enrollment: 14390 (Actual)
Dates: Start 2022-03-14 (Actual); Primary Completion 2025-01-31 (Actual); Study Completion 2025-10-10 (Actual)

PRIMARY OUTCOMES:
Number of participants with higher FNAIT risk characterized by race and ethnicity | At inclusion

SECONDARY OUTCOMES:
Frequency of anti-HPA-1a maternal alloimmunization | At Week 10 postpartum or 10 weeks from the date of pregnancy terminating event
Pregnancy outcomes: incidence of live births, spontaneous abortion, elective abortion, still birth, and premature birth | At Week 10 postpartum or 10 weeks from the date of pregnancy terminating event
Occurrence of neonatal thrombocytopenia | At birth or at the time of the pregnancy terminating event

CONTACTS AND LOCATIONS:
Locations (28):
- United States (19):
  - New Horizons Clinical Trials, LLC, Chandler, Arizona
  - Zillan Clinical Research - Gardena, Gardena, California
  - Yale University School of Medicine, New Haven, Connecticut
  - University of Miami Miller School of Medicine, Miami, Florida
  - Cooper University Hospital, Camden, New Jersey
  - Robert Wood Johnson Medical School, New Brunswick, New Jersey
  - St. Peter's University Hospital, New Brunswick, New Jersey
  - Rutgers New Jersey Medical School, Newark, New Jersey
  - Icahn School of Medicine at Mount Sinai, New York, New York
  - Columbia University Irving Medical Center, New York, New York
  - New York-Presbyterian-Queens, New York, New York
  - Weill Cornell Medicine-New York Presbyterian Hospital, New York, New York
  - University of North Carolina at Chapel Hill, Chapel Hill, North Carolina
  - Ohio State University Wexner Medical Center, Columbus, Ohio
  - Wright State Physicians Obstetrics & Gynecology, Dayton, Ohio
  - Temple Perinatal Diagnosis Center, Philadelphia, Pennsylvania
  - Javara Inc. - Forest, Dallas, Texas
  - The University of Texas Health Science Center at Houston, Houston, Texas
  - Javara Research Inc. - Dallas - PPDS, Houston, Texas
- Sunnybrook Health Sciences Centre, Toronto, Ontario, Canada
- Klinikum der Friedrich Schiller Universität Jena, Jena, Thuringia, Germany
- Leids Universitair Medisch Centrum, Leiden, South Holland, Netherlands
- Norway (2):
  - Oslo Universitetssykehus HF, Ullevål, Oslo, Oslo County
  - Universitetssykehuset Nord Norge, Tromsø
- Sweden (3):
  - Barnmorskestationen Rosengård, Lund, Skåne County
  - Södersjukhuset, Stockholm, Stockholms Ian
  - Clinical Trial Consultants - Uppsala, Uppsala, Uppsala Ian
- St. Thomas' Hospital, London, Surrey, United Kingdom

IPD SHARING:
Plan to Share IPD: No